CLINICAL TRIAL: NCT07208474
Title: The Effect of Laughter Yoga on Burnout and Spiritual Well-Being Among Intensive Care Unit Nurses: A Randomized Controlled Trial
Brief Title: The Effect of Laughter Yoga on Burnout and Spiritual Well-Being
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir Democracy University (Other)
Responsible Party: Principal Investigator, Özüm Erkin, Associate Professor, Izmir Democracy University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IDU-SBE-ÖE-01
Record Dates: First submitted 2025-09-27; First posted 2025-10-06 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Burnout
Keywords: burnout; Spiritual Well-Being
MeSH Terms: conditions — Burnout, Psychological | interventions — Laughter Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- laughter yoga sessions (Experimental): Intervention: Laughter yoga 8 sessions
  Interventions: Other: Laughter yoga
- No Intervention (No Intervention): No Intervention

INTERVENTIONS:
Other: Laughter yoga — Laugher yoga
  Arms: laughter yoga sessions

SUMMARY:
Laughter yoga, a complementary and alternative therapy, is suggested to reduce stress and promote psychological resilience. This study aimed to evaluate the effects of laughter yoga on burnout and spiritual well-being among intensive care nurses.This randomized controlled trial was conducted with 70 intensive care nurses in a university hospital, assigned to the intervention (n = 34) and control (n = 36) groups. The intervention group participated in eight laughter yoga sessions, while the control group received no intervention.

DETAILED DESCRIPTION:
Laughter yoga, a complementary and alternative therapy, is suggested to reduce stress and promote psychological resilience. This study aimed to evaluate the effects of laughter yoga on burnout and spiritual well-being among intensive care nurses.This randomized controlled trial was conducted with 70 intensive care nurses in a university hospital, assigned to the intervention (n = 34) and control (n = 36) groups. The intervention group participated in eight laughter yoga sessions, while the control group received no intervention. Data were collected using the Maslach Burnout Inventory and the Spiritual Well-Being Scale at baseline and after the intervention. Descriptive statistics, paired and independent t-tests, and correlation analyses were performed.

ELIGIBILITY:
Inclusion Criteria: age between 18-65 years, being a ICU nurse, voluntary and at least six months of ICU experience.

-

Exclusion Criteria: prior laughter yoga experience, engagement in other non-pharmacological or pharmacological interventions for burnout, a diagnosed psychiatric disorder requiring medication, physical limitations (e.g., respiratory problems, vertigo, cardiac disease, hernia, epilepsy), recent surgery (within the last three months), lack of internet access or inability to use the online platform, failure to attend all sessions, or incomplete post-test data.

-

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — all genders
Enrollment: 70 (Actual)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2025-07-03 (Actual)

PRIMARY OUTCOMES:
burnout | 1 month
  Maslach Burnout Inventory Scale change from baseline and after the intervention.Maslach Burnout Inventory (MBI) The Maslach Burnout Inventory (MBI), developed by Maslach and Jackson (1981), is designed to assess burnout across three dimensions: emotional exhaustion, depersonalization, and personal accomplishment. The instrument consists of 22 items rated on a five-point Likert scale ranging from 0 (never) to 4 (always). The Turkish adaptation was conducted by Ergin (1992), who modified the original seven-point scale into a five-point format to enhance cultural relevance and interpretability. The subscales include nine items for emotional exhaustion (1, 2, 3, 6, 8, 13, 14, 16, 20), five items for depersonalization (5, 10, 11, 15, 22), and eight items for personal accomplishment (4, 7, 9, 12, 17, 18, 19, 21). Higher scores on the emotional exhaustion and depersonalization subscales, combined with lower scores on the personal accomplishment subscale, indicate greater levels of burnout. T

SECONDARY OUTCOMES:
Spiritual Well-Being | 1 month
  Spiritual Well-Being Scale change from baseline and after the intervention. Spirituality Index of Well-Being (SIWB) The Spirituality Index of Well-Being (SIWB), developed by Daaleman and Frey (2004), is designed to assess individuals' perceptions of their spiritual well-being, with a particular emphasis on meaning and purpose in life. The instrument comprises 12 items rated on a five-point Likert scale ranging from 1 (strongly agree) to 5 (strongly disagree). It includes two subscales: self-efficacy (items 1-7) and life scheme (items 8-12). Total scores range from 12 to 60, with higher scores reflecting greater levels of spiritual well-being.
  The Turkish adaptation was conducted by Serbest and Akgün Şahin (2021), who reported Cronbach's alpha coefficients of 0.858 for the total scale, 0.781 for the self-efficacy subscale, and 0.842 for the life scheme subscale. In the current study, internal consistency was excellent, with Cronbach's alpha coefficients of 0.941 (total), 0.824 (self-ef

CONTACTS AND LOCATIONS:
Locations (1):
- Izmir, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided